CLINICAL TRIAL: NCT05620511
Title: Explore the Neural Mechanism of Mindfulness Training to Reduce Loneliness in Depressed Older Adults: a Randomized Controlled Trial
Brief Title: Explore the Neural Mechanism of Mindfulness Training to Reduce Loneliness in Depressed Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201902151A3
Record Dates: First submitted 2022-11-07; First posted 2022-11-17 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Late Life Depression
Keywords: elderly depression; Mindfulness-based stress reduction (MBSR); MRI; autonomic nervous system
MeSH Terms: interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness based stress reduction (Experimental): 1. Age > 55 years.
  2. Major depressive disorder (MDD).
  3. Right handiness
  4. with a score ≥ 24 on the MMSE
  Interventions: Behavioral: Mindfulness based stress reduction
- Relaxation (Placebo Comparator): 1. Age > 55 years.
  2. Major depressive disorder (MDD).
  3. Right handiness
  4. with a score ≥ 24 on the MMSE
  Interventions: Behavioral: Mindfulness based stress reduction

INTERVENTIONS:
Behavioral: Mindfulness based stress reduction — Mindfulness based stress reduction v.s.Relaxation

SUMMARY:
Perceived loneliness causes a global health burden on older adults. Mindfulness training may be a feasible solution. Through our study, we expect that comprehensive and convincing neuroscientific evidence may support the efficacy underpinning mindfulness training in loneliness reduction.

DETAILED DESCRIPTION:
In this aging and highly industrial society, elderly depression, particularly elderly loneliness, is a growing societal issue. Perceived loneliness not only causes tremendous suffering, disability, cognitive decline, and risk of dementia but also leads to increased mortality. Despite worldwide effort to solve the growing prevalence of loneliness in older adults, no single intervention stands out as universally effective and practical. The exact neural mechanism of loneliness and how the intervention against loneliness takes its effect in the brain remain unclear. Prior studies have indicated that perceived loneliness is associated with distorted cognition toward interpersonal interaction and heightened sympathetic nerve system.Mindfulness training is a discipline that the older adults in our society can readily relate to because the philosophy of mindfulness is similar to Buddhism. Mindfulness trains people to be aware of the surrounding environment and their presence in this environment. Combining the exercises of deep breathing and relaxation, one is taught to be aware of the emotion of oneself to regulate emotion. Mindfulness-based stress reduction (MBSR), a validated and systemized intervention, has been applied to the treatment of depression, anxiety, and insomnia. On the basis of the theory of mindfulness, the investigators estimate that mindfulness can reduce loneliness as well. Thus, the investigators aim to use MBSR in a group of older adults with depression to reduce loneliness. Our previous studies demonstrated that loneliness decreases the grey matter volume in reward system, disrupts the white matter structure, and heightens default-mode network activation. By combining a wearable device for sleep monitoring, heart rate variability measurement, and immune-related cytokine blood test, the investigators can associate these changes with clinical loneliness reduction and brain changes from magnetic resonance imaging. The investigators hope to validate MBSR as an effective intervention against loneliness and explore the supporting neural mechanism.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 55 years.
2. Major depressive disorder (MDD).

Exclusion Criteria:

1. Inability to provide informed consent.
2. Dementia, as defined by MMSE < 24 (<17 if illiterate or no education) and clinical evidence of dementia based on DSM-5 criteria.
3. Lifetime diagnosis of bipolar I or II disorder, schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, or current psychotic symptoms.
4. Abuse of or dependence on alcohol or other substances within the past 3 months, and confirmed by study physician interview.
5. High risk for suicide (e.g., active suicide ideation and/or current/recent intent or plan) AND unable to be managed safely in the clinical trial (e.g., unwilling to be hospitalized). Urgent psychiatric referral will be made in these cases.
6. Non-correctable clinically significant sensory impairment (i.e., cannot hear well enough to cooperate with interview).
7. Unstable medical illness, including delirium, uncontrolled diabetes mellitus, hypertension, hyperlipidemia, or cerebrovascular or cardiovascular risk factors that are not under medical management.
8. Currently under psychotherapy or taking regular meditation or yoga practice (or had experience in these activities)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Loneliness UCLA | Change from Baseline at 3 months
  the severity of loneliness (the score range from 20-80,the lower score means worse)
Mindfulness | Change from Baseline at 3 months
  the effects of mindfulness(the score range from 20-100)
Ham D-17 | Change from Baseline at 3 months
  the insight(the score range from 0-2,the higher score means worse)

SECONDARY OUTCOMES:
Verbal Learning & Memory | Change from Baseline at 3 months
  Word list of Wechsler Memory Scale-III Face memory task(the score range from 0-48,the higher score means better)
structural and functional connectivity | Change from Baseline at 3 months
  Brain MRI connectivity change
Interleukin-1α | Change from Baseline at 3 months
  IL-1α
Interleukin-1β | Change from Baseline at 3 months
  IL-1β
Interleukin-6 | Change from Baseline at 3 months
  IL-6
Interleukin-12 | Change from Baseline at 3 months
  IL-12
TGF-β1 | Change from Baseline at 3 months
  TGF-β1
Total Brain-derived neurotrophic factor | Change from Baseline at 3 months
  Total BDNF
Free Brain-derived neurotrophic factor | Change from Baseline at 3 months
  Free BDNF

CONTACTS AND LOCATIONS:
Locations (1):
- Che-min Lin, Keelung, Taiwan

IPD SHARING:
Plan to Share IPD: No